CLINICAL TRIAL: NCT04056689
Title: A Phase 1b, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL151 in Subjects With Parkinson's Disease
Brief Title: Study to Evaluate DNL151 in Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-C-0003
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Parkinson's Disease
Keywords: LRRK2; Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — DNL151

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- DNL151 Low Dose (Experimental)
  Interventions: Drug: DNL151
- DNL151 Mid Dose (Experimental)
  Interventions: Drug: DNL151
- DNL151 High Dose (Experimental)
  Interventions: Drug: DNL151
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNL151 — Oral repeating dose
  Arms: DNL151 High Dose; DNL151 Low Dose; DNL151 Mid Dose
Drug: Placebo — Oral repeating dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple oral doses of DNL151 in subjects with Parkinson's disease.

DETAILED DESCRIPTION:
This study was previously posted by Denali Therapeutics. In July, 2022, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) between 18 and 35.0 kg/m2, inclusive
* Clinical diagnosis of Parkinson's disease meeting UK Brain Bank criteria and H&Y Stage I, II, or III.
* Able to hold Parkinson's disease medications 8 hours (overnight) prior to specific study assessments

Key Exclusion Criteria:

* Any history of clinically significant asthma, chronic obstructive pulmonary disease, or emphysema within 5 years of screening, or other clinically significant pulmonary disease within 6 months of screening
* Abnormal Vitals including Respiratory Rate, Body Temperature, Blood Pressure, and Pulse Rate
* Pulmonary Function Tests (PFTs) (FVC <60% predicted, FEV1 <50% predicted, FEV1:FVC ratio <0.6, DLCO <70% predicted)
* Clinically significant neurologic disorder other than Parkinson's disease, including history of stroke within 12 months of screening, cognitive impairment, seizure within 5 years of screening, or head trauma with loss of consciousness within 6 months of screening
* Montreal Cognitive Assessment (MoCA) score of <24 at screening

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Randomization to Day 42
Number of Subjects with laboratory test abnormalities | Randomization to Day 42
Number of Subjects with vital sign abnormalities | Randomization to Day 42
Number of Subjects with electrocardiogram (ECG) abnormalities | Randomization to Day 42
Number of Subjects with clinically significant neurological examination abnormalities | Randomization to Day 42

SECONDARY OUTCOMES:
Pharmacokinetic measure of maximum observed plasma concentration (Cmax) of DNL151 | Randomization to Day 28
Pharmacokinetic measure of time to reach maximum observed plasma concentration (Tmax) of DNL151 | Randomization to Day 28
Pharmacokinetic measure of trough plasma observed concentration (Ctrough) of DNL151 | Randomization to Day 28
Pharmacokinetic measure of area under the plasma drug concentration-time curve (AUC) of DNL151 | Randomization to Day 28
Pharmacokinetic measure of CSF concentrations of DNL151 | Randomization to Day 28
Pharmacodynamic measure of pS935 in whole blood | Randomization to Day 28
Pharmacodynamic measure of pRab10 in PBMCs | Randomization to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (8):
- United States (2):
  - PPD Clinical Research Unit, Orlando, Florida
  - Quest Research Institute, Farmington Hills, Michigan
- UZ Leuven, Leuven, Belgium
- Netherlands (2):
  - Centre for Human Drug Research, Leiden, South Holland
  - QPS, Leeuwarden
- United Kingdom (3):
  - Royal Liverpool University Hospital, Liverpool
  - MAC Clinical Research, Manchester
  - Simbec-Orion Clinical Pharmacology, Merthyr Tydfil

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org

REFERENCES:
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102